CLINICAL TRIAL: NCT05191979
Title: Importance of Blood Volume and Its Interaction With Cardiovascular Adaptations
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Copenhagen (Other)
Collaborators: University of Southern Denmark (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: H-21011041
Record Dates: First submitted 2021-12-10; First posted 2022-01-14 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Exercise
Keywords: Blood volume; Cardiac function; Vascular function; Physiological Effects of Long-term exercise training; Mitochondrial function
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Non-blinded, non-randomized intervention design
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blood volume interactions with cardiovascular adaptations (Active Comparator): Individual differences in the time course and relationship between cardiovascular (central and peripheral) adaptations to long-term aerobic training and the concomitant blood volume changes.
  Interventions: Other: Exercise regiment (aerobic exercise on bike)
- Sex differences (Active Comparator): Evaluate differences between genders and hormonal factors influencing individual differences (high vs. low responders) - hypothesizing that female have a blunted cardiovascular response to long-term aerobic training.
  Interventions: Other: Exercise regiment (aerobic exercise on bike)

INTERVENTIONS:
Other: Exercise regiment (aerobic exercise on bike) — Subjects participating in the current study will be trained progressively and intensively for 12 months primarily on bike indoors and outdoors

SUMMARY:
The present project aims to investigate the interaction between training-induced blood volume expansion (plasma- and red blood cell volume responses), central as well as peripheral cardio-vascular adaptations. We will investigate cardiovascular responses through one year of training in recreationally active men and women as well as endurance athletes undertaking shorter training-periods/interventions with environmental heat-stress.

The overall purpose with the project is to investigate the physiological effects of prolonged aerobic exercise on central cardiovascular parameters and peripheral effects in the muscle tissue in untrained individuals. Further, we want to compare these effects to exposure to environmental stress (heat) on performance well trained individuals. The present study consist of three parts using the same methodology in different populations to elucidate the above mentioned mechanisms. The first part is a larger training intervention in untrained/recreationally active men and women aiming at evaluating the initial cardiovascular adaptations to an exercise training regimen. In addition there are two parts aimed to elucidate the mechanisms leading to further improvements in cardiovascular and blood volume adaptations from exercise training in a different environmental condition and artificially elevated PV in already highly adapted endurance athletes.

DETAILED DESCRIPTION:
Background It is well established that a high maximal oxygen consumption (VO2max) is associated with excellent physical performance in endurance sport disciplines. In order to achieve a high V ̇O2max several things must be optimized as according to the Fick equation. One of the main determinants of VO2max is the oxygen carrying capacity of the blood, which is dictated by the total hemoglobin mass and is significantly higher in endurance athletes than untrained individuals.

Naturally, this system is tightly regulated to maintain a steady blood composition and to promptly recover blood volume if lost due to i.e. hemorrhage but can also be altered by exercise and or exposure to extreme environmental conditions. Changes in blood volume and composition can be seen already after two weeks of conventional exercise training where increases in PV are seen in combination with elevated erythropoietin (EPO) while red blood cell volume remains unaffected. This supports the proposed notion of the kidney acting as a "critmeter" and that a reduced hematocrit due to expansion of PV thereby may regulate erythropoiesis. In already trained individuals i.e. athletes, PV and Hbmass can be further increased through repeated and or prolonged exposure to altitude or hot environmental conditions.

Research questions and hypothesis

1. Explore gender and individual differences in the time course and relationship between cardiovascular (central and peripheral) adaptations to long-term aerobic training and the concomitant blood volume changes.
2. Evaluate differences between genders and factors influencing individual differences (high vs. low responders) - hypothesizing that female have a blunted cardiovascular response to long-term aerobic training.
3. What is the relative significance of blood volume, muscle metabolic and cardiovascular adaptations for performance and aerobic power.

An incremental exercise test on a cycle ergometer will be conducted to determine the maximal work rate and VO2max. Four venous blood samples, each 4 ml, is taken during the rest period. Subjects blood volume and body composition are evaluated with a DXA-scan and CO-rebreathing technique after a brief period of rest following the exercise test.

In the second experimental trials (visit 2), participants will be familiarized to the experimental protocol by cycling in the semi-recumbent position. For the experiment participants will undergo a standardized test of orthostatic tolerance by a lower-body negative pressure (LBNP) of -15mmHg for maximally 10 min and -30mmHg for maximally 10 min. Ventricular function are measured at both levels of LBNP. After the orthostatic tolerance test the subject will perform semi-recumbent cycling at two submaximal intensities with euhydration (control). At least 30 min after the first bout of exercise (after the subject have returned to baseline hemodynamic levels), subjects will ingest a hypertonic beverage with the aim of increasing PV by ~15% (intervention). Ventricular function is again measured before the second bout of semi-recumbent submaximal cycling is initiated at the same intensities as before mentioned.

In the third visit (visit 3) we will measure whether the exercise regimen have effects on peripheral (arm) blood flow regulation. The peripheral vascular function is determined by measures of brachial artery diameter and blood velocity using duplex ultrasonography before and after flow-mediated dilation (FMD) where a cuff positioned around the upper arm is inflated to 200 mmHg for 5 min for then to be deflated. Vascular sensitivity and endothelial function is then measured by ultrasound before and after infusion of the vasoactive drugs Acetylcholine (Ach) (25 and 100 μg min-1 (kg arm-mass)-1), Sodium Nitroprusside (SNP) (0.75, 1.5 and 3.0 μmol min-1 L arm-mass-1). Between all these measurements there will be a break of minimum 15 min. Before the subject leaves this visit for the first time (baseline) two muscle biopsy's of approximately 150 mg is also taken for cultivation of cells and assessment of changes in capillary density, muscle fiber composition and mitochondrial density and function. One muscle biopsy will also be taken during visit one at sampling point after 2 weeks, 1, 2 and 6 months after baseline and with two muscle biopsy's at 12 months after the baseline round making for a total of eight biopsy's for each subject.

After the first round of experiment has concluded the subjects will undergo an exercise regimen for 12 months, consisting of 3-4 supervised and monitored cycling training sessions weekly. The exercise training will be supervised and structured in a progressive manner to accustom the subjects to regular and high intensity exercise. Subjects will again undergo study procedures at 2 weeks 1, 2, 6, and 12 months after baseline measures in order to allow for continuous analysis of the short- and long-term cardiovascular adaptations. In addition we want to measure coronary blood flow, muscle mitochondrial volume - and function to determine the effects of central versus peripheral adaptations to long term training at baseline, 2, 6 and 12 months.

In order to discern any central cardiovascular effects from peripheral we want to acutely normalize blood volume by phlebotomy at the final visit of the 12 month exercise training. Before and after phlebotomy, VO2max and Q̇max will be determined to investigate any central cardiovascular adaptations.

Subjects in this project are subjected to the following measures: Cardiac and vascular ultrasound, muscle biopsies, Catheterization with arterial and venous blood samples, CO-rebreathing technique, DXA-scan, Electrocardiogram (ECG), Flow-mediated dilation, vasodilator response to intra-arterial infusion of Ach and SNP, LBNP, performance test, and Phlebotomy.

ELIGIBILITY:
Inclusion Criteria:

* absence of metabolic, chronic diseases, uncontrolled arrhythmia, 2. or 3. degree AV-block or sick sinus syndrome
* no history of smoking or alcohol consumption (≥ 14 items / week)
* decent acoustic window for echocardiography.

Exclusion Criteria:

* chronic disease or taking medication
* history of >2 years of exercise training
* failure to meet exercise raining criteria

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-01-06 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Maximal systemic oxygen uptake | 20 minutes
  Training-induced changes in maximal systemic oxygen uptake (ml/min) is evaluated with an incremental maximal cycle protocol on a cycle ergometer
Resting and cycling stroke volume and function measured with echocardiography | 90 minutes
  LV stroke volume (ml) and LV basal and apical twist (Deg) will be used to measure training-induced changes in LV function during exercise
Change in vascular conductance of the brachial artery | 2 hours
  Assessment of changes in arm vascular conductance (ml/min/mm/Hg/kg arm mass) to flow mediated dilation, infusion of Acetylcholine and sodium nitroprusside, assessed by ultrasound Doppler.
Blood volume | 20 minutes
  Training-induced changes in total blood volume (mL) is measured using the Carbon-monoxide rebreathing method.

SECONDARY OUTCOMES:
Mitochondrial biogenesis | 60 minutes
  Expression of complex I-V will be analyzed in order to evaluate if the applied training induced mitochondrial biogenesis.
Fat mass | 20 minutes
  Training-induced changes in fat mass (kg) is determined by dual-energy x-ray absorptiometry (DXA)-scan
Fat free mass | 20 minutes
  Training-induced changes in fat free mass (kg) is determined by DXA-scan
Cardiac dimentions | 90 minutes
  Changes in left ventricular linear dimensions and left ventricular mass; left ventricular volumes; left ventricular ejection fraction; left atrial size; right heart parameters are determined by echocardiography during rest

CONTACTS AND LOCATIONS:
Overall Officials: Nikolai B. Nordsborg, Prof., Principal Investigator — University of Copenhagen - Department of Nutrition, Exercise and Sports
Locations (2):
- Denmark (2):
  - Department of Nutrition, Exercise and Sports, Copenhagen
  - University of Copenhagen, Copenhagen

IPD SHARING:
Plan to Share IPD: Undecided
Fully anonymous data will be shared with other researchers.